CLINICAL TRIAL: NCT06594653
Title: Evaluation of Outcomes Related to Walking in a Rehabilitation Program Supported by Robotics (Lokomat) in Children Suffering from Congenital and Acquired Brain Injuries
Brief Title: Evaluation of Outcomes of Robotics Rehabilitation in Cerebral Palsy
Acronym: LK
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: ID 1123
Record Dates: First submitted 2024-08-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy; Gait Disorders, Neurologic
Keywords: Robotic Rehabilitation; Gait
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: pre treatment assesment — All measurements will be obtained using an optoelectronic multicamera system for human motion analysis (with eight high-resolution cameras with infrared light and a sampling frequency of 60 Hz. The experimental protocol requires the positioning of markers (plastic spheres covered by reflecting film, 10 mm in diameter). Markers will be placed by clinical operators (physiotherapists with training in optoelectronic system for human motion analysis) after training and experience in recognition of the position of body landmarks.
Other: post treatment assessment — All measurements will be obtained using an optoelectronic multicamera system for human motion analysis (with eight high-resolution cameras with infrared light and a sampling frequency of 60 Hz. The experimental protocol requires the positioning of markers (plastic spheres covered by reflecting film, 10 mm in diameter). Markers will be placed by clinical operators (physiotherapists with training in optoelectronic system for human motion analysis) after training and experience in recognition of the position of body landmarks.

SUMMARY:
The use of robotic devices in rehabilitation programs can improve walking patterns by reorganizing joint kinematics. This study aims to quantify the effects of a rehabilitation program supported by the Lokomat (Hocoma) robotic device on walking in children and young people with movement disorders, considering different levels of impairment.

DETAILED DESCRIPTION:
Cerebral Palsy is one of the most common neuromotor disorders in pediatric age, characterized by permanent movement and posture impairments, often affecting walking. In recent decades, advancements in robotics have revolutionized rehabilitation. Studies have shown that combining conventional physiotherapy with robotic rehabilitation tools offers greater benefits in patient recovery. At the IRCCS Eugenio Medea, a robotic rehabilitation program using the Lokomat (Hocoma) has been implemented for several years to improve walking in children and young people with walking disorders. The investigators hypothesize that robotic devices can enhance walking ability (e.g., speed, stride length) and reorganize joint kinematics. This study aims to quantify the effects of this treatment based on the level of impairment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CP;
* able to walk independently with or without assistance

Exclusion Criteria:

* presence of behavioral problems;
* presence of uncontrolled seizures
* presence of severe visual disturbances.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The subjects enrolled in the present study are patients diagnosed with infantile cerebral palsy, able to walk independently with or without assistance. The subjects enrolled are patients who have been regularly hospitalized at the IRCCS Medea to carry out a rehabilitation program with the aid of Lokomat. Patients with behavioral problems, uncontrolled seizures, severe visual disturbances, multiple muscle-tendon retraction pattern, painful symptoms upon mobilization of the lower limbs are excluded.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the rehabilitation program in terms of gait speed | Through study completion, an average of 1 year
  Starting from the data collected through Gait Analysis for each subject during the pre-treatment and post-treatment sessions, the walking speed [m\s] will be calculated. Moreover, the pre- and post-treatment results will be compared for each subject.
Effectiveness of the rehabilitation program in terms of cadence | Through study completion, an average of 1 year
  Starting from the data collected through Gait Analysis for each subject during the pre-treatment and post-treatment sessions, the walking cadence [step/min] will be calculated. Moreover, the pre- and post-treatment results will be compared for each subject.
Effectiveness of the rehabilitation program in terms of stride length | Through study completion, an average of 1 year
  Starting from the data collected through Gait Analysis for each subject during the pre-treatment and post-treatment sessions, the stride length [mm] will be calculated. Moreover, the pre- and post-treatment results will be compared for each subject.
Effectiveness of the rehabilitation program in terms of step width | Through study completion, an average of 1 year
  Starting from the data collected through Gait Analysis for each subject during the pre-treatment and post-treatment sessions, the step width [mm] will be calculated. Moreover, the pre- and post-treatment results will be compared for each subject.
Effectiveness of the rehabilitation program in terms of gait phase | Through study completion, an average of 1 year
  Starting from the data collected through Gait Analysis for each subject during the pre-treatment and post-treatment sessions, the gait phase [cycle%] will be calculated. Moreover, the pre- and post-treatment results will be compared for each subject.
Effectiveness of the rehabilitation program in terms of lower limbs ROM | Through study completion, an average of 1 year
  Starting from the data collected through Gait Analysis for each subject during the pre-treatment and post-treatment sessions, the lower limbs ROM [°] will be calculated. Moreover, the pre- and post-treatment results will be compared for each subject.
Effectiveness of the rehabilitation program in terms of summary gait parameters GDI | Through study completion, an average of 1 year
  Starting from the data collected through Gait Analysis for each subject during the pre-Starting from the data collected through Gait Analysis for each subject during the pre-treatment and post-treatment sessions, the summary gait parameter Gait Deviation Index (GDI) will be calculated. A GDI of 100 or higher indicates the absence of gait pathology. Moreover, the pre- and post-treatment results will be compared for each subject.
Effectiveness of the rehabilitation program in terms of summary gait parameters GPS | Through study completion, an average of 1 year
  Starting from the data collected through Gait Analysis for each subject during the pre-Starting from the data collected through Gait Analysis for each subject during the pre-treatment and post-treatment sessions, the summary gait parameter Gait Profile score (GPS)[°] will be calculated. A GPS of 7 or lower indicates the absence of gait pathology. Moreover, the pre- and post-treatment results will be compared for each subject.

SECONDARY OUTCOMES:
Treatment effect based on the level of impairment about walk fatique | Through study completion, an average of 1 year
  For each subject, we administered the 6-Minute Walking Test to define impairment levels (moderate vs. severe impairment). The improvement of each group will be evaluated.(moderate vs. severe impairment). The improvement of differn group will be evaluate.
Treatment effect based on the level of impairment about gross motor ability | Through study completion, an average of 1 year
  For each subject, we administered the Gross Motor Function Classification System (GMFCS) to define impairment levels, distinguishing between moderate and severe impairments. The GMFCS consists of five levels: Level I indicates no walking impairment, while the subsequent levels indicate increasing degrees of impairment. The improvement of each group (moderate vs. severe impairment) will be evaluated.
Treatment effect based on the level of impairment about functional activity | Through study completion, an average of 1 year
  For each subject, we administered the Functional Activities Questionnaire (FAQ) to define impairment levels, distinguishing between moderate and severe impairments. FAQ sum scores range from 0 to 30, with a cut-off of 9 indicating dependence in three or more activities. The improvement of each group (moderate vs. severe impairment) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Piccinini, Principal Investigator — Istituto di Ricovero e Cura a Carattere Scientifico Eugenio Medea
Locations (1):
- IRCCS E. Medea, Bosisio Parini, Italy, Italy

IPD SHARING:
Plan to Share IPD: No